CLINICAL TRIAL: NCT03179163
Title: Peripheral Vascular Effects of Sulfhydryl-containing Antihypertensive Pharmacotherapy on Microvascular Function and Vessel Remodeling in Hypertensive Humans
Brief Title: Peripheral Vascular Effects of Sulfhydryl-containing Antihypertensive Pharmacotherapy on Microvessels in Humans
Acronym: H2SPharm
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: COVID shut down human subjects research and then the grant funding expired
Sponsor: Penn State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lacy Alexander, Associate Professor Kinesiology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY3224; 5R01HL093238 (NIH); 120058 (Other: FDA)
Record Dates: First submitted 2017-06-02; First posted 2017-06-07 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hypertension,Essential
Keywords: Hypertension; Blood Pressure; Cardiovascular Disease; Angiotensin Converting Enzyme (ACE) Inhibitor; Diuretic; Nitric Oxide; Hydrogen Sulfide; Captopril; Enalapril; Hydrochlorothiazide; Microcirculation; Skin
MeSH Terms: conditions — Essential Hypertension; Hypertension; Cardiovascular Diseases | interventions — Captopril; Enalapril; Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: Subjects are grouped as normal (<120/80 mmHg) and hypertensive (≥140/90 mmHg and <160/110 mmHg). All subjects undergo one round of experiments. Hypertensive subjects received randomly-assigned antihypertension medication angiotensin converting enzyme inhibitor with a sulfahydrl donor (ACEi+SH), angiotensin converting enzyme inhibitor (ACEi), or diuretic for 16 weeks and then repeat experiments. Normotensive subjects receive no intervention and repeat experiments16 weeks after initial experiments as a time control.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Outcomes Assessor are masked according to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Normotensive (No Intervention): Blood Pressure <120/80 mmHg
- Hypertensive - ACE inhibitor with sulfahydrl donor (ACEi +SH) (Experimental): Captopril Pill intervention Blood Pressure ≥140/90 mmHg and <160/110 mmHg
  Interventions: Drug: Captopril Pill
- Hypertensive - ACE inhibitor (ACEi) (Experimental): Enalapril Pill intervention Blood Pressure ≥140/90 mmHg and <160/110 mmHg
  Interventions: Drug: Enalapril Pill
- Hypertensive - Diuretic (Active Comparator): Hydrochlorothiazide intervention Blood Pressure ≥140/90 mmHg and <160/110 mmHg
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Captopril Pill — ACEi+SH
  Other Names: National Drug Code (NDC) # 00781-8061-01
  Arms: Hypertensive - ACE inhibitor with sulfahydrl donor (ACEi +SH)
Drug: Enalapril Pill — ACEi
  Other Names: NDC# 51672-4039-03
  Arms: Hypertensive - ACE inhibitor (ACEi)
Drug: Hydrochlorothiazide — diuretic
  Other Names: NDC# 00603-3857-32
  Arms: Hypertensive - Diuretic

SUMMARY:
High blood pressure can cause physical changes to the blood vessels of the body (remodeling). If a person who has high blood pressure also has a lot of blood vessel remodeling with their condition, they are more likely to have poor results with medical treatment for hypertension. The researchers examine the impact of different classes of drugs that doctors use to treat high blood pressure (hypertension) on blood vessel remodeling. Some drugs that doctors prescribe for their patients contain a "sulfhydryl group" (a sulfur atom bonded to a hydrogen atom). Drugs that have the sulfhydryl group may reduce blood vessel remodeling more that drugs that do not. For this study, participants who have high blood pressure perform the experiments, take a drug for 16-weeks to lower blood pressure, and repeat the experiments. The researchers randomly assign one of three drugs to participants who have high blood pressure: a diuretic ("water pill"), a drug containing a sulfhydryl (SH) group, or a drug that does not contain a sulfhydryl group. Participants who do not have high blood pressure perform the experiments, but do not take any of the drugs. In some of our experiments, the researchers use a technique called "microdialysis" (MD). With MD, the researchers perfuse some research drugs into the skin on the forearm through tiny tubing that mimics capillaries. These MD drugs mimic or block substances the body naturally makes to control the small blood vessels in the skin. The drugs remain in nickel-sized areas around the tubing and do not go into the rest of the body. The researchers also analyze very small skin samples (skin biopsy) obtained from the forearm. Lastly, the researchers use a standard technique called "flow mediated dilation" (FMD) that uses blood pressure cuffs and ultrasound to look at the health of larger blood vessels in the body. FMD includes placing a small tablet of nitroglycerin under the tongue during part of the test.

DETAILED DESCRIPTION:
Upon initial screening and again within a week of testing, all subjects will have an assessment of 24-hour ambulatory blood pressure. Subject screening will be performed by the Penn State Clinical Translational Research Center (CTRC) medical staff and will include a physical exam by a clinician, anthropometry, and a chemical and lipid profile, liver and renal function. Women will be either postmenopausal (absence of menstruation of >1 year and Follicle Stimulating Hormone (FSH) >25 milli-international units per milliliter (mlU/ml)) and not be taking hormone replacement therapy, or normally menstruating and tested in the early follicular phase of their cycle. Subjects will also go through an assessment of conduit vessel endothelial and vascular smooth muscle function with brachial artery flow-mediated vasodilation (FMD), and sublingual nitroglycerin.

Subjects will undergo initial microdialysis experiments and biopsy samples will be obtained. Subjects will then be randomly assigned to treatment group. Blood pressure will be monitored every 2 weeks and weekly compliance checks will be made by the researcher's nurse coordinator. 24-hour ambulatory blood pressure monitoring will be conducted monthly to determine the efficacy of antihypertensive treatment and to inform dosing titration. Examining pharmacokinetic and dynamic data from the literature indicate that blood pressure lowing and peripheral vascular effects are maximized by 12 weeks of antihypertensive therapy and maintained thereafter. After 16 weeks of the assigned intervention, subjects will repeat microdialysis experiments and additional cutaneous biopsy samples will be obtained. Conduit artery measures including brachial artery FMD and responsiveness to sublingual nitroglycerin will also be evaluated at this time.

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* 40-65 years
* Blood pressure: Normotensive <120/80 mmHg Hypertensive ≥140/90 mmHg and <160/110 mmHg
* HbA1C of <6.5%
* Women are post-menopausal and not taking hormone replacement therapy, or have normal cycles and are tested in the early follicular phase
* Subjects may or may not be taking one doctor-prescribed drug to lower blood pressure (e.g. diuretic, ACE inhibitor).

  * Must be able to stop physician-prescribed antihypertensive drug for the duration of the subject's participation in the study (with the approval of their personal physician).

Exclusion Criteria:

Relevant to all subjects:

* current medications which could conceivably alter the cardiovascular or thermoregulatory control or responses (e.g. beta blockers, calcium channel blockers, ACE inhibitors, angiotensin receptor blockers)
* taking a diuretic (also see below)
* allergy to test substances
* allergy to latex
* nicotine use (smoking, chewing tobacco, etc.)
* illegal/recreational drug use
* pregnancy or breastfeeding
* diabetes

Relevant to hypertensive subjects only:

* contraindication for all three pharmacotherapy drugs used in this study

  o Note: Subjects who have a contraindication (e.g. a condition, medication with a known interaction, known allergy) to only one or two of the three pharmacotherapy drugs, may be assigned one of the pharmacotherapy drugs that is not contraindicated.
* history of having taken an ACE inhibitor with antioxidant properties (e.g. Captopril, Zofenopril)
* kidney problems
* liver problems
* history of heart disease or failure
* history of blood clots or stroke
* angioedema
* electrolyte imbalance
* planned surgery requiring general anesthesia during the pharmacotherapy period
* peripheral vascular disease
* diuretics (a subject taking only a diuretic to control the subject's hypertension may be included in the study if the subject stops taking the diuretic for the duration of the subject's participation in the study with the approval of the subject's personal physician.)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lacy M Alexander, PhD, Principal Investigator — Penn State University
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recuited out of the Centre County region and had Stage II hypertension based on resting seated brachial blood pressure. Other than hypertension, all participants were clinically healthy.
Groups:
- Hypertensive - ACEi +SH: Captopril Pill intervention Blood Pressure ≥140/90 mmHg and <160/110 mmHg
  Captopril Pill: ACEi+SH
Period: Overall Study
Arm/Group | Hypertensive - ACEi +SH
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hypertensive - Sulfahydrdryl-donaging ACE Inhibitor: Captopril Pill intervention Blood Pressure ≥140/90 mmHg and <160/110 mmHg
  Captopril Pill 50-100 mg twice daily
Arm/Group | Hypertensive - Sulfahydrdryl-donaging ACE Inhibitor
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Endothelium Dependent Vasodilation
Description: This measurement is performed using a laser Doppler flow meter. The flow meter produces a non-invasive qualitative and dimensionless index of blood flow in blood vessels during the localized perfusion of the endothelium-dependent vasodilatory acetycholine in a dose response fashion. The results are the differences in the area under the curve units=(laser Doppler flux/MAP)*logAch concentration
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: (flux/MAP)*logAch (mol/L)
Arm/Group | Hypertensive - ACEi +SH
Number analyzed (Participants) | 10
(flux/MAP)*logAch (mol/L) | 83 (47)
Statistical Analysis 1: Comparison: Hypertensive - ACEi +SH; A priori power analysis (power = 0.80,a= 0.05) confirmed a sample size of n= 10 was needed to determine a meaningful difference of 10% in the (flux/MAP)*logAch(mol/L) . All data were analyzed with repeated-measures ANOVA . When appropriate, post hoc Tukey-Kramer corrections were applied to correct for multiple comparisons. Significance was set a priori at a<0.05; Test type: Other; p = 0.01, ANOVA; Mean Difference (Net) = 0.01

2. Secondary Outcome: Systolic Blood Pressure
Description: Blood pressure is measured via brachial auscultation manually or with a critical care monitor. The peak blood pressure during a cardiac cycle when the heart contracts.
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hypertensive - ACEi +SH
Number analyzed (Participants) | 10
mmHg | 122 (8)

3. Secondary Outcome: Diastolic Blood Pressure
Description: Blood pressure is measured via brachial auscultation manually or with a critical care monitor. The lowest blood pressure during a cardiac cycle when the heart is between beats.
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hypertensive - ACEi +SH
Number analyzed (Participants) | 10
mmHg | 80 (8)

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Hypertensive - ACEi +SH
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT03179163/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT03179163/ICF_001.pdf